CLINICAL TRIAL: NCT03742752
Title: Enteral Versus Parenteral Nutrition in the Conservative Treatment of Upper Gastrointestinal Fistula After Surgery: a Multicenter, Randomized, Parallel-group, Open Label
Brief Title: Enteral Versus Parenteral Nutrition in the Conservative Treatment of Upper Gastrointestinal Fistula After Surgery
Acronym: NUTRILEAK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: default inclusion
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016_74; 2018-A01625-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-10-29; First posted 2018-11-15 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2020-09

CONDITIONS: Gastrointestinal Fistula; Enteral Nutritional Support
Keywords: enteral nutrition; parenteral nutrition; gastrointestinal fistula
MeSH Terms: conditions — Digestive System Fistula; Hyperphagia | interventions — Enteral Nutrition; Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral Nutrition (EN) (Experimental): To demonstrate the superiority of EN versus TPN in the treatment of postoperative upper GI anastomotic leak (PUGIAL) after upper GI surgery (including esophageal, gastric, duodenal, pancreatic and obesity surgery).
  Patients will be randomized to receive EN through jejunostomy or nasojejunal tube until oral diet covering at least 60% of their daily requirement
  Interventions: Other: Enteral nutrition
- Parenteral Nutrition (TPN) (Active Comparator): Patients will be randomized to receive TPN through central venous access, piccline or totally implantable venous access port tube until oral diet covering at least 60% of their daily requirement
  Interventions: Other: Parenteral nutrition

INTERVENTIONS:
Other: Enteral nutrition — administration of enteral nutrition
  Arms: Enteral Nutrition (EN)
Other: Parenteral nutrition — administration of parenteral nutrition
  Arms: Parenteral Nutrition (TPN)

SUMMARY:
The incidence of clinically significant anastomotic leaks (AL) after upper gastrointestinal (GI) surgery is approximately 4 % - 20 %, and the associated mortality can be as high as 80 % . Nutritional support is a key component of therapy in such cases, related to high prevalence of malnutrition and nil per month required for leak treatment.

In the prophylactic setting, before the occurrence of any AL, a literature review based on seven randomised trials showed that enteral nutrition (EN) is associated with shorter hospital stay, lower incidence of severe of infectious complications, lower severity of complications and decreased cost compared to parenteral nutrition (TPN) following major upper GI surgery .

In the curative setting, after the AL occurrence, very few evidence is available. Only one randomized clinical trial suggested the superiority of EN versus TPN after pancreatic surgery with a increase of the 30-day fistula closure rate from 37% in the TPN group to 60% in the EN group .

This sole randomised study available did not include all postoperative upper GI AL (PUGIAL) that can occur after esophageal, gastric, duodenal, pancreatic surgery (including obesity surgery), whereas the concept of enteral nutritional support is highly relevant for all these situations.

However surgeons are usually reluctant to provide EN in case of AL. A randomized study suggested the feasibility of EN in 47 patients with upper GI AL but no randomized study to date has been designed to test the superiority of EN versus TPN in PUGIAL.

The study aim is to demonstrate the superiority of EN versus TPN to accelerate AL healing after upper GI surgery.

Hypothesis:

EN increases the 30-day fistula closure rate in PUGIAL, allowing better HRQOL without increasing morbi-mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Patients having received upper GI surgery for benign or malignant disease including, oesophageal, gastric, duodenal or pancreatic surgery or bariatric surgery
* Diagnosis of an active postoperative fistula or persisting after a failure of surgical or endoscopic procedure dedicated to close the fistula
* AL diagnosed from less than 72h AND confirmed on at least two criteria among the followings:
* clinical symptoms of AL
* ct scan / ultrason imaging and /or endoscopic diagnosis of AL
* biologic/bacteriology diagnosis on fluid output
* intraoperative diagnosis of AL at time of reoperation
* Indication of nil per mouth
* American society of anesthesiologist score 1, 2 or 3
* In case of neoplasm, absence of peritoneal carcinomatosis or distant metastasis
* No severe concomitant uncontrolled disease
* Life expectancy more than 6 months
* No history of allergy or study product intolerance
* Ongoing healthcare insurance

Exclusion Criteria:

* - Scheduled surgical or endoscopic treatment with the aim to close the fistula (suture, prosthesis, clip or glue). In case of such treatment failure, patients are eligible to participate to the study. Endoscopic or surgical drainage are not exclusion criteria (meaning that drainage only is authorized before randomization)
* History of or current severe uncontrolled cardiovascular, pulmonary, renal or liver failure
* Uncontrolled sepsis related to the AL
* Malnutrition requiring combined nutritional treatment with the enteral AND parenteral routes together
* Untreated or persistent Peritoneal carcinomatosis or distant metastasis
* Pregnant and/or lactating women
* Freedom privacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
30-day fistula closure rate | 30 days after randomization
  Fistula closure will be defined as an output of no fluid for at least 48 hours in wound or drainage AND absence of any fluid collection on imaging (Computed Tomography scan with injection of contrast product).

SECONDARY OUTCOMES:
6-month fistula closure rate | at 6 months after randomization
  Percentage of patients having their fistula closed according to the definition above within 6 months after randomization
Time to first fistula closure | at 6 months after randomization
  Time to first fistula closure defined as time in days from randomization to first AL closure within 6 months after randomization
Treatment-related complications | longitudinal evaluation during all the study duration (from randomization to 6 months)
  number of patients presenting at least one complication related to the nutritional support (catheter related infection or thrombosis, tube related complication)
Postoperative mortality rate | at 30 days after randomization
  rate of death after operation
Postoperative morbidity rate | at 30 days after randomization
  rate of patients with a Clavien-Dindo grade 3-4-5 complications
Weight | longitudinal evaluation during all the study duration (from randomization to 6 months)
  in kg
Albumin and prealbumin | longitudinal evaluation during all the study duration (from randomization to 6 months)
  in g/L
C reactive protein | longitudinal evaluation during all the study duration (from randomization to 6 months)
  mg/L
Grip test | longitudinal evaluation during all the study duration (from randomization to 6 months)
  muscular strength
Length of hospital stay in healthcare structure | from the randomization until the end of hospitalization, up to 6 months
  Length of hospital stay in healthcare structure (including home hospitalization) based on the number of days of hospitalization
Short form questionnaire 36 (SF-36) | at inclusion, day 30, day 60, 3 months and 6 months
  Patient's Health-related quality of life (HRQOL) score. The SF-36 includes a single-item measure of health transition or change. he SF-36® Health Survey items and scales were constructed using the Likert method of summated ratings.4 Answers to each question are scored (some items need to be recoded). These scores are then summed to produce raw scale scores for each health concept which are then transformed to a 0 - 100 scale. Thie higher the score is, the better the quality of life is.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Piessen, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France

REFERENCES:
- [Derived] Gronnier C, Chambrier C, Duhamel A, Dervaux B, Collet D, Vaudoyer D, Regimbeau JM, Jougon J, Thereaux J, Lebreton G, Veziant J, Valverde A, Ortega-Deballon P, Pattou F, Mathonnet M, Perinel J, Beyer-Berjot L, Fuks D, Rouanet P, Lefevre JH, Cattan P, Deguelte S, Meunier B, Tuech JJ, Pessaux P, Carrere N, Salame E, Benaim E, Dousset B, Msika S, Mariette C, Piessen G; FRENCH association. Enteral versus parenteral nutrition in the conservative treatment of upper gastrointestinal fistula after surgery: a multicenter, randomized, parallel-group, open-label, phase III study (NUTRILEAK study). Trials. 2020 Jun 2;21(1):448. doi: 10.1186/s13063-020-04366-3. PMID 32487210